CLINICAL TRIAL: NCT01774370
Title: A Regulatory Requirement Non-interventional Study to Monitor the Safety and Effectiveness of Pradaxa (Dabigatran Etexilate Mesilate, 110 mg or 150 mg b.i.d.) in Korean Patients With Non-valvular Atrial Fibrillation(SPARK: Safety Study of Pradaxa in AF Patients by Regulatory Requirement of Korea)
Brief Title: SPARK: Safety Study of Pradaxa in Atrial Fibrillation Patients by Regulatory Requirement of Korea
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.139
Record Dates: First submitted 2013-01-16; First posted 2013-01-24 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2018-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pradaxa group
  Interventions: Drug: Pradaxa (Dabigatran etexilate mesilate)

INTERVENTIONS:
Drug: Pradaxa (Dabigatran etexilate mesilate) — 110 mg or 150 mg b.i.d.

SUMMARY:
This is a prospective, non-interventional, open-label, multi-centre study. It will provide additional safety information of Pradaxa in Korean patients with non-valvular AF in clinical settings.

DETAILED DESCRIPTION:
Study Design:

regulatory Post Marketed Surveillance study

ELIGIBILITY:
Inclusion criteria:

* Age >= 18 years at enrollment
* Patients who have been started on Pradaxa in accordance with the approved label in Korea
* Patients who have signed on the data release consent form

Exclusion criteria:

* Patients with previous exposure to Pradaxa
* Clinically significant bleeding
* Increased risk of bleeding due to following diseases;

  * Recent gastrointestinal ulceration
  * Recent intracranial or intracerebral bleeding history
  * Intraspinal or intracerebral vascular abnormalities
  * Recent brain, spinal or ophthalmic surgery
  * Recent brain or spinal injury
  * Known or suspected oesophageal varices
  * Arteriovenous malformations
  * Vascular aneurysms
  * Presence of malignant neoplasms at high risk of bleeding
* Concomitant treatment with any other anticoagulants e.g. unfractionated heparin (UFH), low molecular weight heparins (enoxaparin, dalteparin etc), heparin derivatives (fondaparinux etc), oral anticoagulants (warfarin, rivaroxaban, apixaban etc) except under the circumstances of switching therapy to or from Pradaxa or when UFH is given at doses necessary to maintain an open central venous or arterial catheter
* Severe renal impairment (CrCl < 30mL/min)
* Concomitant treatment with oral ketoconazole or dronedarone
* Patients hypersensitive to dabigatran or dabigatran etexilate or to any ingredient in the formulation
* Prosthetic heart valve replacement
* No creatinine clearance collected within at least one year prior to enrollment
* Current participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with non-valvular AF
Sampling Method: Probability Sample
Enrollment: 3182 (Actual)
Dates: Start 2013-01-14 (Actual); Primary Completion 2017-02-17 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is a prospective, non-interventional, open-label, multi-centre study.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended a specialist sites which ensured that they met all strictly implemented inclusion/exclusion criteria. Subjects were not to be entered to trial treatment if any one of the specific entry criteria was violated.
Groups:
- Pradaxa Group: Physician carefully reviewed the special precautions for use in patients with risk of bleeding before determining the dose of Pradaxa and patients were prescribed dabigatran dose for 24±2 weeks from the options described below:
  * Dabigatran etexilate mesilate 110 mg b.i.d. (oral administration of one capsule twice daily )
  * Dabigatran etexilate mesilate 150 mg b.i.d. (oral administration of one capsule twice daily)
Period: Overall Study
Arm/Group | Pradaxa Group
Started | 3182
Completed | 3053
Not Completed | 129
Not completed — Never taken the PRADAXA during the study | 4
Not completed — Administered prior to the contract date | 4
Not completed — Subjects of contraindications | 34
Not completed — Violated inclusion/exclusion criteria | 53
Not completed — Follow-up failure | 34

BASELINE CHARACTERISTICS:
Population: Safety analyses will be based on all patients treated, i.e. all patients who received at least one dose of Pradaxa.
Arm/Group | Pradaxa Group
Number analyzed (Participants) | 3053
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.26 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1201
  Male | 1852
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Adverse Events(Including Unexpected Adverse Events, Serious Adverse Events, Drug-related Adverse Events, Adverse Events Leading to Discontinuation and Adverse Events by Intensity, Outcome of the Event, Causality)
Description: Occurrence of adverse events(Including unexpected adverse events, serious adverse events, drug-related adverse events, adverse events leading to discontinuation and adverse events by intensity, outcome of the event, causality).
  Number analyzed presents the "Number of participants with Adverse events"
Time Frame: up to 26 weeks
Population: Safety analyses will be based on all patients treated, i.e. all patients who received at least one dose of Pradaxa.
Measure: Number; unit: Adverse events
Arm/Group | Pradaxa Group
Number analyzed (Participants) | 672
Adverse events | 871

2. Secondary Outcome: Percentage of Participants With Stroke
Description: Stroke was defined as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of haemorrhage or infarction.
Time Frame: up to 26 weeks
Population: Effectiveness Analysis set: Effectiveness analysis will be performed to the patients who have been on Pradaxa more than 12 weeks (in case of long-term follow up, 24 weeks).
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa Group
Number analyzed (Participants) | 2311
percentage of participants
  Yes: number analyzed (Participants) | 7
  Yes | 0.30
  No: number analyzed (Participants) | 2304
  No | 99.70

3. Secondary Outcome: Percentage of Participants With Systemic Embolism
Description: Systemic embolism was defined as an acute vascular occlusion of the extremities or any organ (kidneys, mesenteric arteries, spleen, retina or grafts) and was to be documented by angiography, surgery, scintigraphy or autopsy.
Time Frame: up to 26 weeks
Population: Effectiveness Analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Pradaxa Group
Number analyzed (Participants) | 2311
percentage of participants
  Yes: number analyzed (Participants) | 0
  No | 100.0

ADVERSE EVENTS:
Time Frame: All adverse events occurring from the start of Pradaxa treatment up to 7 days after last follow-up visit; up to 26 weeks
Arm/Group | Pradaxa Group
All-Cause Mortality (participants affected / at risk) | 5/3053
Serious Adverse Events (participants affected / at risk) | 104/3053
Other Adverse Events (participants affected / at risk) | 0/3053
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pradaxa Group (N=3053)
Dyspepsia (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 3
Gastric ulcer (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 11
Transient ischaemic attack (Nervous system disorders) | 7
Cerebrovascular accident (Nervous system disorders) | 4
Dementia (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Dizziness postural (Nervous system disorders) | 1
Brain stem infarction (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Chest discomfort (General disorders) | 1
Asthenia (General disorders) | 1
Oedema (General disorders) | 1
Death (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Atrial fibrillation (Cardiac disorders) | 6
Atrial flutter (Cardiac disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Mitral valve disease mixed (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Cellulitis (Infections and infestations) | 3
Pneumonia (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Clonorchiasis (Infections and infestations) | 1
Encephalitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Haematuria (Renal and urinary disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Hypotension (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 2
Aortic aneurysm (Vascular disorders) | 1
Arterial rupture (Vascular disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Radiation proctitis (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Subarachnoid hemorrhage (Injury, poisoning and procedural complications) | 1
Cataract (Eye disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Alcoholic liver disease (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-10): https://cdn.clinicaltrials.gov/large-docs/70/NCT01774370/Prot_SAP_000.pdf